CLINICAL TRIAL: NCT02675582
Title: Investigation of the Acute Calming Effects of Drinks Containing Herbal Extracts in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Collaborators: Northumbria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1509
Record Dates: First submitted 2016-01-21; First posted 2016-02-05 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Cognitive Function and Mood

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): Mix 1 flavored still beverage
  Interventions: Other: Herbal Beverage
- Herbal beverage 1 (Experimental): Mix 2 flavored still beverage with a botanical extract(1)
  Interventions: Other: Herbal Beverage
- Herbal Beverage 2 (Experimental): Mix 3 flavored still beverage with a botanical extract(2)
  Interventions: Other: Herbal Beverage
- Combined Herbal Beverage (Experimental): Mix 4 flavored still beverage with 2 botanical extracts (1,2)
  Interventions: Other: Herbal Beverage

INTERVENTIONS:
Other: Herbal Beverage — Intervention involves consuming one beverage at the beginning of each visit during the incomplete block design sequence

SUMMARY:
The primary objectives of this study are to assess the effects of three investigational drinks containing three botanicals in differing combinations versus a placebo control, on mood, psychological state, physical response, and cognitive performance during and after exposure to an observed multi-tasking stressor.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 49 years
* Self-report of good health
* Are not excluded on the basis of the following exclusion criteria

Exclusion Criteria:

* Are a smoker
* Have food allergies or sensitivities to any of the ingredients contained in the investigational product or any other foodstuff
* Currently take medication except the contraceptive pill
* Have habitually used dietary supplements within the last month (defined as more than 3 consecutive days or 4 days in total)
* Have sleep disturbances and/or are taking sleep aid medication Are employed in a job that includes night shift work
* Have a Body Mass Index (BMI) outside of the range 18-35 kg/m2or weigh less than 50kg or more than 85kg.
* Have high blood pressure (systolic over 139 mm Hg or diastolic over 89 mm Hg)
* Have a history of neurological, vascular or psychiatric illness including epilepsy or seizures (excluding depressive illness and anxiety)
* Have a history of anxiety or a current diagnosis of anxiety or depression
* Are pregnant, trying to get pregnant or breast feeding
* Have a recent history of (within 12 months of screening visit) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as more than 60g (men) / 40g (women) pure alcohol per day (7 / 5.5 units)
* Have learning difficulties or dyslexia
* Have visual impairment that cannot be corrected with glasses or contact lenses
* Have frequent migraines that require medication (more than or equal to 1 per month)
* Have disorders of the blood (e.g. anaemia, hemophilia, thrombocytosis)
* Have a heart disorder or a history of vascular illness
* Have a respiratory disorder that requires regular medication (Note: participants with asthma who only take their medication occasionally/as required are eligible for this study)
* Have a diagnosis of type I or type II diabetes
* Have a history of renal or hepatic disease, or other severe diseases of the gastrointestinal tract (e.g. iron accumulation, iron utilization disorders, hypercalcaemia, hypercalciuria), that are likely to interfere with metabolism/absorption/secretion of the product under investigation
* Have any health condition that would prevent fulfillment of the study requirements
* Are currently or have in the past 8weeks participated in other clinical or nutrition intervention studies
* Have participated in the BPNRC's recent stress study
* Do not have a bank account (required for payment)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in mood | Pre dose, 60, 150, 240 min post dose
  During each assessment mood and psychological state will be assessed before and after performance of an observed multi-tasking stressor via completion of the 'State' subscale of the State-Trait Anxiety Inventory and computerised versions of the Bond-Lader visual analogue mood scales and separate visual analogue scales (VAS) measuring subjective stress, relaxation and calmness.

SECONDARY OUTCOMES:
Change in Cognitive function | Pre dose, 60, 150, 240 min post dose
  During each assessment mood and psychological state will be assessed before and after performance of an observed multi-tasking stressor via completion of the 'State' subscale of the State-Trait Anxiety Inventory and computerised versions of the Bond-Lader visual analogue mood scales and separate visual analogue scales (VAS) measuring subjective stress, relaxation and calmness.

CONTACTS AND LOCATIONS:
Overall Officials: David Kennedy, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided